CLINICAL TRIAL: NCT03003858
Title: Retrospective Observational Trial on the Role of a Hyaluronic Acid Medical Device in Pediatric Patients Affected by Gingivitis
Brief Title: Hyaluronic Acid and Gingivitis in Pediatrics
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Other Study IDs: IDS DipCh 04
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Gingivitis
Keywords: gingivitis; hyaluronic acid; pediatrics; medical devices
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: 0.1% HA-based film-forming device (Gengigel Prof® Fluid) — 0.1% HA-based film-forming device (Gengigel Prof® Fluid, Ricerfarma, Milano, Italy) administered (oral rinses for 3-5 min.) three to five times a day over a 4-week period as an adjunct to domiciliary care and oral hygiene instructions and motivation

SUMMARY:
The purpose of this observational, non-controlled, single site trial with a retrospective design is to verify, in a large paediatric population affected by gingivitis, the tolerability and safety of 0.1% HA-based film-forming devices (Gengigel Prof® Fluid, Ricerfarma) administered three to five times a day over a 4-week period as an adjunct to domiciliary care and oral hygiene instructions

DETAILED DESCRIPTION:
The efficacy and safety data belonging to clinical trials with Hyaluronic Acid (HA) in oral mucosa pathologies (gingivitis, post-surgical treatment of incisions of the buccal cavity, periodontitis and other pathological periodontal conditions) have been confirmed in about 20 years of clinical practice by dentists. Starting from this experience, several clinical centers, including our institute, have been introducing over the last years HAbased film-forming devices in pediatrics. In particular, we have been using a liquid formulation with 0.1% HA; it has been routinely administered in our clinic during the routine pre-visit by Nurses and Dental Hygienist to children with gingivitis and given to the parents to administered to the children in the post visit period as an adjunct to domiciliary care and oral hygiene instructions. The product we used is featured by the following additional characteristics:

* a high concentration of HA, which explains its efficacy in reducing swelling and secondary pain;
* a liquid formulation, which can easily treat the whole gingival area, including the points of more difficult access;
* and at last, a really acceptable taste, that plays an interesting role to obtain a good compliance from young patients.

The variables collected in this observational trial are the same collected during our current clinical practice: Gingival Index (GI), Plaque Index (PII), Bleeding on probing (BOP), count of edematous gingival sites and AE/SAE for safety.

ELIGIBILITY:
Inclusion Criteria:

* Any gender and age between 6 and 16 years
* healthy condition and with a clinical diagnosis of mild to moderate gingivitis
* Gingival Index (GI) from 1 to 2 (0= Normal gingiva; 1= Mild inflammation - slight change in color and slight edema but no bleeding on probing; 2= Moderate inflammation - redness, edema and glazing, bleeding on probing; 3= Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding)
* Plaque Index (PII) over then 7% (0= no plaque; 1= a film of plaque adhering to the free gingival margin, adjacent to the tooth; 2= moderate accumulation of soft deposits within the gingival pocket or between the tooth and gingival margin; 3= abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin)
* Bleeding on probing (BOP) over then 5%

Exclusion Criteria:

* taking antibiotics or anti-inflammatory drugs during or for 1 month prior to the study.
* any relevant systemic disease which is known to cause gingivitis
* history of any allergic reaction to HA
* to treat the gingivitis with any other medication/mouthwashes in the period of the study.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with a clinical diagnosis of mild to moderate gingivitis with at least 3 of the following:
  * red, swollen, and spongy gums;
  * gums that bleed spontaneously or after brushing, eating or touching;
  * having bad breath;
  * sensation of tingling or itching of the gums;
  * presence of pus in the pockets between teeth.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
tolerability of 0.1% HA-based film-forming device | 4 week
  tolerability of 0.1% HA-based film-forming devices (Gengigel Prof® Fluid, Ricerfarma) administered three to five times a day over a 4-week period as an adjunct to domiciliary care and oral hygiene instructions

CONTACTS AND LOCATIONS:
Overall Officials: Gianpietro Farronato, MD, Principal Investigator — Dipartimento di Scienze Chirurgiche, Ricostruttive e Diagnostiche, IRCCS Cà Granda Ospedale Maggiore Policlinico, Milano, (Italy); Marco Tremolati, Investigator, Study Director — ASP Istituto Pio Albergo Trivulzio, Milano (Italy)

IPD SHARING:
Plan to Share IPD: Yes